CLINICAL TRIAL: NCT03195010
Title: Management of Venous Thromboembolic Events (VTE) in Patients With Hematologic Disorders and Treatment-Induced Thrombocytopenia: A Pilot Study
Brief Title: Management of Platelet Transfusion Therapy in Patients With Blood Cancer or Treatment-Induced Thrombocytopenia
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Terminated because of slow recruitment and lack of funding support
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 9799; NCI-2017-00864 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 9799 (Other: Fred Hutch/University of Washington Cancer Consortium); P30CA015704 (NIH)
Record Dates: First submitted 2017-06-13; First posted 2017-06-22 (Actual); Results first posted 2019-10-21 (Actual); Last update posted 2019-10-21 (Actual); Status verified 2019-10

CONDITIONS: Acute Biphenotypic Leukemia; Acute Lymphoblastic Leukemia; Acute Myeloid Leukemia; B-Cell Non-Hodgkin Lymphoma; Chronic Lymphocytic Leukemia; Chronic Myelogenous Leukemia, BCR-ABL1 Positive; Hematologic and Lymphocytic Disorder; Hematopoietic Cell Transplantation Recipient; Myelodysplastic Syndrome; Primary Myelofibrosis; Secondary Myelofibrosis; T-Cell Non-Hodgkin Lymphoma; Thrombocytopenia; Venous Thromboembolism
MeSH Terms: conditions — Leukemia, Biphenotypic, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Lymphoma, B-Cell; Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Hematologic Diseases; Myelodysplastic Syndromes; Primary Myelofibrosis; Lymphoma, T-Cell; Thrombocytopenia; Venous Thromboembolism | interventions — Platelet Transfusion

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group I (lower dose platelet transfusion) (Experimental): Patients undergo platelet transfusion on all days when the morning platelet count is below the threshold 30 x 10^9/L for up to 30 days or until the platelet count spontaneously recovers to > 50 x 10^9 for 3 consecutive days in the absence of transfusions.
  Interventions: Biological: Platelet Transfusion
- Group II (higher dose platelet transfusion) (Experimental): Patients undergo platelet transfusion on all days when the morning platelet count is below the threshold 50 x 10^9/L for up to 30 days or until the platelet count spontaneously recovers to > 50 x 10^9 for 3 consecutive days in the absence of transfusions.
  Interventions: Biological: Platelet Transfusion

INTERVENTIONS:
Biological: Platelet Transfusion — Undergo lower dose platelet transfusion
  Other Names: Blood Platelet Transfusion
  Arms: Group I (lower dose platelet transfusion)
Biological: Platelet Transfusion — Undergo higher dose platelet transfusion
  Other Names: Blood Platelet Transfusion
  Arms: Group II (higher dose platelet transfusion)

SUMMARY:
This pilot clinical trial compares the safety of two different platelet transfusion "thresholds" among patients with blood cancer or treatment-induced thrombocytopenia whose condition requires anticoagulant medication (blood thinners) for blood clots. Giving relatively fewer platelet transfusions may reduce the side effects of frequent platelet transfusions without leading to undue bleeding.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine feasibility of a randomized controlled trial comparing two different platelet transfusion thresholds (50 x 10^9/L versus [vs] 30 x 10^9/L) in patients with treatment or malignancy-induced thrombocytopenia requiring therapeutic anticoagulation.

SECONDARY OBJECTIVES:

I. Progressive or new venous thromboembolic (VTE).

II. Progressive or new arterial thromboembolism (ATE).

III. Hemorrhagic events (World Health Organization [WHO] grade 2 or greater).

IV. A composite of I, II and III.

V. Major bleeds (WHO grade 3 or 4).

VI. Number of platelet transfusions per patient during the study period.

VII. Platelet transfusion related complications (including transfusion reactions, alloimmunization and volume overload).

VIII. Degree to which platelet target thresholds are achieved.

OUTLINE: Patients are randomized into 1 of 2 groups.

GROUP I (Lower dose): Patients undergo platelet transfusion on all days when the morning platelet count is below the threshold 30 x 10^9/L for up to 30 days or until the platelet count spontaneously recovers to > 50 x 10^9 for 3 consecutive days in the absence of transfusions.

GROUP II (Higher dose): Patients undergo platelet transfusion on all days when the morning platelet count is below the threshold 50 x 10^9/L for up to 30 days or until the platelet count spontaneously recovers to > 50 x 10^9 for 3 consecutive days in the absence of transfusions.

After completion of study, patients are followed up at 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Any patient with non-acute promyelocytic leukemia (APL) acute leukemia (acute myeloid leukemia [AML], acute lymphoblastic leukemia [ALL], biphenotypic leukemia) undergoing curative intent chemotherapy OR any patient undergoing allogeneic hematopoietic stem cell transplantation (HSCT) for a hematologic disorder (including acute leukemia as above, chronic myelogenous leukemia [CML], chronic lymphocytic leukemia [CLL], myelodysplastic syndrome [MDS], primary or secondary myelofibrosis, hypereosinophilic syndromes, plasma cell disorders, B-cell or T-cell lymphoma)
* Disease may be measurable or non-measurable
* Diagnosis of symptomatic venous thromboembolism requiring therapeutic-dose anticoagulation (unfractionated or low-molecular weight heparin or oral anticoagulants) throughout the period of hematopoietic recovery
* Anticipated platelet count =< 50 x 10^9/L for >= 5 days within 72 hours of enrollment
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Separate episode of VTE or arterial thrombosis within 3 months of enrollment
* Major bleed (WHO grade 3 or 4) within 6 months of enrollment
* Active bleeding (grade 2 or higher) at the time of enrollment
* History of intracranial bleeding at any time
* Disorders of hemostasis including von Willebrand disease, hemophilia, platelet function disorders
* Concomitant use of aspirin or non-steroidal anti-inflammatory drugs
* Evidence of disseminated intravascular anticoagulation (DIC) as determined by the patient's primary provider
* History of alloimmunization (defined as platelet refractoriness with panel reactive antibody [PRA] > 25%) at the time of or prior to enrollment
* Uncontrolled or concurrent illness including, but not limited to, ongoing or active infection, unstable angina pectoris
* Psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant or able to become pregnant and unwilling to use two forms of birth control during the study period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2017-06-09 (Actual); Primary Completion 2018-12-21 (Actual); Study Completion 2018-12-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Garcia, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Group I (Lower Dose Platelet Transfusion) | Group II (Higher Dose Platelet Transfusion)
Started | 2 | 2
Completed | 2 | 2
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group I (Lower Dose Platelet Transfusion) | Group II (Higher Dose Platelet Transfusion) | Total
Number analyzed (Participants) | 2 | 2 | 4
Age, Continuous [Mean (Full Range); unit: years] | 42 [23 to 61] | 35 [30 to 40] | 39 [23 to 61]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 2 | 4
Region of Enrollment [Number; unit: participants]
  United States | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Number of Eligible Patients Approached for the Study
Time Frame: Up to 1 year
Measure: Count of Participants; unit: Participants
Groups:
- Approached Patients: Eligible patients approached for participation
Arm/Group | Approached Patients
Number analyzed (Participants) | 4
Participants | 4

2. Primary Outcome: Number of Patients Approached for But Refusing Consent
Description: Reasons for ineligibility will be reported qualitatively in order to inform future studies.
Time Frame: Up to 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Approached Patients
Number analyzed (Participants) | 4
Participants | 0

3. Primary Outcome: Number of Patients Consenting to Enrollment
Time Frame: Up to 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Approached Patients
Number analyzed (Participants) | 4
Participants | 4

4. Primary Outcome: Number of Patients Eligible
Time Frame: Up to 1 year
Measure: Count of Participants; unit: Participants
Groups:
- Screened Patients: Patients screened for eligibility
Arm/Group | Screened Patients
Number analyzed (Participants) | 7
Participants | 4

5. Primary Outcome: Number of Patients Screened and Deemed Ineligible
Description: Reasons for ineligibility will be reported qualitatively in order to inform future studies.
Time Frame: Up to 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Screened Patients
Number analyzed (Participants) | 7
Participants | 3

6. Primary Outcome: Number of Patients Successfully Following Protocol
Description: Will evaluate the number of patients successfully following protocol, defined as receiving transfusions 'on protocol' at the end of the study period.
Time Frame: Up to 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Group I (Lower Dose Platelet Transfusion) | Group II (Higher Dose Platelet Transfusion)
Number analyzed (Participants) | 2 | 2
Participants | 2 | 2

7. Secondary Outcome: Incidence of Hemorrhagic Events (World Health Organization Grade 2 or Greater)
Description: Will evaluate the incidence of hemorrhagic events (World Health Organization grade 2 or greater).
Time Frame: Up to 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Group I (Lower Dose Platelet Transfusion) | Group II (Higher Dose Platelet Transfusion)
Number analyzed (Participants) | 2 | 2
Participants | 0 | 0

8. Secondary Outcome: Major Bleeds (World Health Organization Grade 3 or 4)
Description: Will evaluate the major bleeds (World Health Organization grade 3 or 4).
Time Frame: Up to 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Group I (Lower Dose Platelet Transfusion) | Group II (Higher Dose Platelet Transfusion)
Number analyzed (Participants) | 2 | 2
Participants | 0 | 0

9. Secondary Outcome: Number of Platelet Transfusions Per Patient During the Study Period
Time Frame: Up to 1 year
Measure: Mean (Full Range); unit: platelet transfusions
Arm/Group | Group I (Lower Dose Platelet Transfusion) | Group II (Higher Dose Platelet Transfusion)
Number analyzed (Participants) | 2 | 2
platelet transfusions | 2 [2 to 2] | 9 [5 to 13]

10. Secondary Outcome: Percent of Days on Which Subjects Are Transfused (or Transfusion Are Not Given)
Description: The frequency with which transfusions are given despite a platelet count above the determined threshold will be documented, as will the frequency with which transfusions are not administered within 24 hours after a platelet count below the determined threshold.
Time Frame: Up to 1 year
Measure: Number; unit: percentage of study days
Arm/Group | Group I (Lower Dose Platelet Transfusion) | Group II (Higher Dose Platelet Transfusion)
Number analyzed (Participants) | 2 | 2
percentage of study days | 0 | 3.8

11. Secondary Outcome: Platelet Transfusion Related Complications
Description: Total number of transfusion reactions, patients experiencing alloimmunization and volume overload will be reported.
Time Frame: Up to 1 year
Measure: Number; unit: Platelet transfusion complication
Arm/Group | Group I (Lower Dose Platelet Transfusion) | Group II (Higher Dose Platelet Transfusion)
Number analyzed (Participants) | 2 | 2
Platelet transfusion complication | 0 | 2

12. Secondary Outcome: Progressive or New Arterial Thromboembolism
Description: Will evaluate the progression or new arterial thromboembolism by either documented acute electrocardiographic changes compatible with myocardial injury and/or serum biochemical changes diagnostic of myocardial infarction, or documented imaging (computed tomography or magnetic resonance imaging) changes compatible with infarct due to embolism in the presence of a new neurological deficit, or imaging demonstrated intraluminal filling defects in an arterial distribution accompanied by symptoms of acute ischemia (acute onset pain, pallor, loss of pulses or other end-organ damage).
Time Frame: Up to 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Group I (Lower Dose Platelet Transfusion) | Group II (Higher Dose Platelet Transfusion)
Number analyzed (Participants) | 2 | 2
Participants | 0 | 0

13. Secondary Outcome: Progressive or New Venous Thromboembolic
Description: Will evaluate the progressive or new venous thromboembolic. Will require imaging confirmation, defined as intraluminal filling defect(s) on contrast-enhanced computed tomography or incompressible venous segment(s) on ultrasonography.
Time Frame: Up to 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Group I (Lower Dose Platelet Transfusion) | Group II (Higher Dose Platelet Transfusion)
Number analyzed (Participants) | 2 | 2
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: On study time (varied between subjects)
Arm/Group | Group I (Lower Dose Platelet Transfusion) | Group II (Higher Dose Platelet Transfusion)
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/2
Other Adverse Events (participants affected / at risk) | 1/2 | 2/2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group I (Lower Dose Platelet Transfusion) (N=2) | Group II (Higher Dose Platelet Transfusion) (N=2)
mucositis (Gastrointestinal disorders) | 1 (1) | 2 (2) — Related to chemotherapy
transaminitis (Gastrointestinal disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-12-27): https://cdn.clinicaltrials.gov/large-docs/10/NCT03195010/Prot_SAP_000.pdf